CLINICAL TRIAL: NCT02169687
Title: Pilot, Monocentric, Non-comparative Study of the Effectiveness and Safety of High Intensity Focused Ultrasound Device in Patients With Autonomous Hyperfunctioning Thyroid Nodules
Brief Title: High Intensity Focused Ultrasound Device in Patients With Autonomous Hyperfunctioning Thyroid Nodules
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Protocol's modifications requested by IRB weren't feasible to continue the study
Sponsor: Theraclion (Industry)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other); Hôpital Saint Louis Paris (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU/F/02.01/Protocol V0
Record Dates: First submitted 2014-05-05; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Autonomous Hyperfunctioning Thyroid Nodules
Keywords: Thyroid, HIFU, hyperfunctioning, autonomous
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hifu (Experimental)
  Interventions: Device: HIFU

INTERVENTIONS:
Device: HIFU — High Intensity focalized Ultrasounds

SUMMARY:
The purpose of this study is to assess the efficacy and safety of High Intensity Focalized Ultrasound (HIFU) in the treatment for toxic Thyroids nodules

DETAILED DESCRIPTION:
Hyperthyroidism is defined by a decrease in thyrotropin (TSH) level associated with elevated or normal free T4 and T3 (subclinical hyperthyroidism). The most frequent etiology in the older population is toxic adenoma or toxic multinodular goiter. Several studies have demonstrated that such hyperthyroid status was associated with an increase in cardiac arrhythmias (atrial fibrillation) and an increase in cardiovascular mortality. Nevertheless, the management of patients presenting with subclinical hyperthyroidism remains controversial.

Surgery is indicated in case of large toxic adenomas especially in young patients. In European countries, radioiodine treatment is indicated in older patients, especially presenting with cardiothyreosis or when surgery is contraindicated. Radioiodine is a simple, cost-effective, and safe procedure in the treatment of autonomously hyperfunctioning thyroid nodule. In a prospective study [Nygaard, 1999], there was a 45% decrease in the total thyroid volume within 3 months after radio-iodine treatment, and 75% of patients with no previous anti-thyroid drug treatment normalized for thyroid function within 3 months. In another recently published prospective study [Endorgan, 2004], there was a decrease in hot nodules volume assessed by US of 28.8% 3 months, 46.2% 6 months and 54% 12 months after radioiodine treatment, and 66.7% of patients were euthyroid at 3 months, 71.8% at 6 months, 76.9% at 12 months. The AACE guidelines for the diagnosis and management of thyroid nodules [Feld, 1996] recommend that all patients with toxic autonomous thyroid nodules require treatment and remind that radioactive iodine is the treatment of choice for most patients with toxic nodules. Nevertheless, at the present time there are no published data that demonstrate the effectiveness of radioiodine treatment on the prevention of cardiac complications in case of subclinical hyperthyroidism. When radioiodine treatment is proposed, physicians must follow regulations and policies on 131I in Europe and US. The European Union recently adopted the main international commission on radiological protection (ICRP) recommendations on radiation protection. Such regulation may raise a number of practical problems for 131I treated patients. With the exception of a few countries as Germany and Switzerland, there often is no legislation defining the maximal dose of radioiodine that can be administered on an ambulatory basis. Policies and recommendations have been proposed to reduce the radiation hazards for the public or the family leaving around the radioiodine treated patients.

Therefore, because of these radioprotection recommendations, and because of contraindication to surgery and to radioiodine in some cases, an alternative treatment for toxic nodular nodules, HIFU, may be suggested.

The aim of the study is to assess the efficacy and safety of HIFU treatment for autonomous hyperfunctioning thyroid nodules. The main objective of the study is to assess the rate of patients with TSH normalization (or increase). US changes of treated nodules, especially the nodule volume, will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, aged at least 18 years.
* Patient presenting with at least one autonomous hyperfunctioning thyroid nodule

  * TSH 0,1 mU/ml
  * Hyperfunctioning at thyroid scintigraphy with partial or total extinction of parenchyma
* Targeted nodules visible with ultrasonography
* Volume to be treated 15 cc
* Targeted area located at least at 2 mm from the trachea, the esophagus, and the carotid artery.
* Composition of the targeted nodule: no more than 75% cystic.
* Absence of abnormality at laryngoscopy in recurrent nerves
* Voluntary consent (patient or legal guardian) to participate in the study, following a full explanation of the nature and purpose of the study, by signing the Informed Consent document at the eligibility assessment visit
* Patients for whom iodine therapy is contra-indicated or unfeasible and surgery is contra-indicated or refused
* Patients refusing iodine therapy
* Willingness and availability to return for all required follow-up visits and to undergo all required study procedures.
* Patient affiliated to the French Health Insurance System

Exclusion Criteria:

* For the targeted nodule(s): presence of signs evidencing a nodule malignancy (compression or curvature of the surrounding organs, positive or suspicious previous FNAB).
* Suspicious cervical lymph nodes at US
* > 75% Cystic nodule
* Macrocalcification inducing a shadow in the thyroid significant enough to preclude the HIFU treatment
* Pregnant or lactating woman. Female patient of childbearing age will be screened for pregnancy prior to enrollment in the study and will be included only if having a suitable contraception method.
* Known latex or lidocaine hypersensitivity
* History of neck irradiation or subtotal thyroidectomy
* Non controlled evolutive cardiothyreosis
* Patients treated with antithyroid medications within the month before the pre-treatment visit
* Subjects whose concurrent illnesses, disability, or geographical residence would hamper regular attendance at required study visits
* Patients who have received any investigational drug or device within the last 30 days and/or patients who are currently participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patient with TSH normalization / increase | 3 months

SECONDARY OUTCOMES:
Number of patients with TSH normalization / increase | 3 weeks, 6 months, 12 months
Changes of FT3 and FT4 | D3, D14, 6 weeks, M3, M6, M12
Change in the volume nodule | 6 weeks, M3, M6 and M12
Number of adverse events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié Salpetrière, Paris, Paris, France